CLINICAL TRIAL: NCT02478086
Title: Effects of High vs. Standard Protein Intake in the Weight Gain and Renal Function Security in Newborn Extreme Premature
Brief Title: Effects of High vs. Standard Protein Intake in Newborn Extreme Premature
Acronym: experimental
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Collaborators: Instituto Mexicano del Seguro Social (Other Government); Universidad de Guanajuato (Other)
Responsible Party: Principal Investigator, Guadalupe Gómez Rodríguez, Guadalupe Gómez Rodríguez Médico neonatologo, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R-2012-1002-63
Record Dates: First submitted 2015-05-31; First posted 2015-06-23 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Abnormal Renal Function; Malnutrition
Keywords: amino acids; renal function; extreme premature
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- use amine acids parenteral 3.5g (Experimental): Amino acids parenteral (Levamin Nomo 10% ®) Group A with an initial doses of amino acids until reaching 3.5 g/kg/day during 28 days.For the study of renal function baseline urea, creatinine and BUN were measured within 24 h after birth in order to avoid any alteration cost by mother alter kidney function, afterwards the same markers were measured at the day 7, 14, 21 and 28. These markers were measure using orto-clinical diagnostic series 50-0278 USA.
  The anthropometric measurements were assessed weekly by the same person to avoid bias (cephalic perimeter and height); weight was measured weekly using the same scale (SECA model 3741321009, Germany). All anthropometric and lab results were kept in a collection sheet.
  Interventions: Dietary Supplement: use amine acids parenteral 3.5g
- use amine acids parenteral 4g (Experimental): Group B with an initial doses of 2.5 g/kg/day with daily increments of 0.5 g/kg/day until reaching 4 g/kg/day during 34 days.Weight, urea, creatinine and blood urea nitrogen (BUN) were measured weeklyFor the study of renal function baseline urea, creatinine and BUN were measured within 24 h after birth in order to avoid any alteration cost by mother alter kidney function, afterwards the same markers were measured at the day 7, 14, 21 and 28. These markers were measure using orto-clinical diagnostic series 50-0278 USA.
  The anthropometric measurements were assessed weekly by the same person to avoid bias (cephalic perimeter and height); weight was measured weekly using the same scale (SECA model 3741321009, Germany). All anthropometric and lab results were kept in a collection sheet.
  Interventions: Dietary Supplement: use amine acids parenteral 4g

INTERVENTIONS:
Dietary Supplement: use amine acids parenteral 3.5g — Group A we administered standard doses of amino acids was administered (3.5gr) the study of renal function baseline urea, creatinine and BUN were measured within 24 h after birth in order to avoid any alteration cost by mother alter kidney function, afterwards the same markers were measured at the day 7, 14, 21 and 28. These markers were measure using orto-clinical diagnostic series 50-0278 USA.
  The anthropometric measurements were assessed weekly by the same person to avoid bias (cephalic perimeter and height); weight was measured weekly using the same scale (SECA model 3741321009, Germany). All anthropometric and lab results were kept in a collection sheet.
  Other Names: Levamin Nomo 10% 3.5g / kg / day
  Arms: use amine acids parenteral 3.5g
Dietary Supplement: use amine acids parenteral 4g — Group B we administered high doses of amino acids was administered (4 gr) the study of renal function baseline urea, creatinine and BUN were measured within 24 h after birth in order to avoid any alteration cost by mother alter kidney function, afterwards the same markers were measured at the day 7, 14, 21 and 28. These markers were measure using orto-clinical diagnostic series 50-0278 USA.
  The anthropometric measurements were assessed weekly by the same person to avoid bias (cephalic perimeter and height); weight was measured weekly using the same scale (SECA model 3741321009, Germany). All anthropometric and lab results were kept in a collection sheet.
  Other Names: Levamin Nomo 10% 4g / kg / day
  Arms: use amine acids parenteral 4g

SUMMARY:
Introduction:

The preterm newborn of extremely low birth weight (PNELW), endures adverse nutritional conditions to mimic intrauterine growth. It´s known that amino acids contribute to protein synthesis, but also intervene in weight gain. Most newborns receive amino acids throw parenteral nutrition at a doses of 3.5gr/k/day, that doses its unable to reach the birth weight when discharged, so the weight its below the 10th percentile, which rises the risk for presenting alterations in neurodevelopment.

Objective:

To compare a higher doses of parenteral amino acids vs. standard doses, expecting an increased weight gain in the high amino acid doses group, meanwhile following the renal function security profile

Methods:

A randomize, single blind clinical trial, carried on, in the Neonatology Service of Unidad Medica de Alta Especialidad Numero 48 of the Instituto Mexicano del Seguro Social, in the city of Leon, Mexico. Between the period of 1st August 2012 to 31 January 2013. A standard doses of amino acids was administered (3.5gr) to a control group and a high doses (4gr) to an experimental group. Weight, urea, creatinine and blood urea nitrogen (BUN) were measured weekly. In the study were included all preterm newborns (PN) weighting less than 1500 grs and with less than 32 weeks of gestational age that match all the inclusion criteria. Statics Analysis: descriptive statistics were calculates, also chi2 test and Fisher Exact test were applied to categorical variables, t-student test to continuous variables, and ANOVA in multiple groups.

DETAILED DESCRIPTION:
METHODS:

Types of study: randomized single-blinded clinical trial. Time and place of development: Neonatology Service (NICU, Neonatal Ward and Premature Ward) in the Unidad Medica de Alta Especialidad Número 48, of Instituto Mexican del Seguro Social in Leon, Mexico, in the period between 1st of August 2012 and 31st of January 2013. This study was approved by local ethical committees of the hospital and University of Guanajuato. Informed consent was requested in writing to parents to include their children into the study

Inclusion Criteria

1. Preterm infant of less than 32 gestational weeks and weighting less than 1500g.

Exclusion criteria

1. Preterm infant with severe congenital malformation
2. Patients with acute kidney failure.
3. Inform consent form not signed.

Methodology For the accomplishment of the present trial all premature patients weighting less than 1500g and less than 32 weeks of age were included, and also the patients referred by the other units in less than 24h after birth. Randomization was carried out using closed envelopes with the assigned amino acid doses, constituting two groups: group A with an initial doses of 2.5 g/kg/day with daily increments of 0.5 g/kg/day until reaching 3.5 g/kg/day; group B with an initial doses of 2.5 g/kg/day with daily increments of 0.5 g/kg/day until reaching 4 g/kg/day.

The amino acids administered are from Pisa Laboratory (Levamin Nomo 10%, ®), with the following composition in every 100 ml: 511 mg of L-isoleucine, 725mg of L-leucine, 934 mg of L-licina, 396 mg of L-methionine, 724 mg of L-phenylalanine, 514 of L-threonine, 180mg of L-tryptophan, 668 mg of L-valine, 1025 mg of L-arginine, 443 mg of L-histidine, 1469 mg of L-alanine, 40 mg of L-Sistine, 1198 mg of Glycine, 590 mg of L-proline, 500 mg of L-serine, 235 mg of L-aspartic acid, 309 mg of L-glutamine acid and 36mg of L-tyrosine.

For the study of renal function baseline urea, creatinine and BUN were measured within 24 h after birth in order to avoid any alteration cost by mother alter kidney function, afterwards the same markers were measured at the day 7, 14, 21 and 28. These markers were measure using orto-clinical diagnostic series 50-0278 USA.

The anthropometric measurements were assessed weekly by the same person to avoid bias (cephalic perimeter and height); weight was measured weekly using the same scale (SECA model 3741321009, Germany). All anthropometric and lab results were kept in a collection sheet.

The presence of sepsis was diagnosed using clinical signs of systemic inflammatory response and a positive blood culture, necrotizing enterocolitis was diagnosed using Bell's criteria and permeable artery duct was defined by a connection between the aorta and the pulmonary artery with a left to right shunt; death was also evaluated.

Sample Size The sample size was calculated for 24 patients in each group as necessary to detect a delta of 15% in the weight variable (beta error of 20 % and alpha error of 5%). 10% losses were assumed, resulting in a total of 28 needed patients per group.

Statistical analysis

Central tendency measures were used for all variables and also chi square test for qualitative variables were applied, T-student test for continuous variables ad for multiple measurements ANOVA Test was applied. The software used was NCSS v. 8.0 (Kaysville, Utah USA)

ELIGIBILITY:
Inclusion Criteria:

1. Preterm infant of less than 32 gestational weeks and weighting less than 1500g

Exclusion Criteria:

1. Preterm infant with severe congenital malformations.
2. Patients with acute kidney failure.
3. Inform consent form not signed.

Ages: 1 Day to 4 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2012-08; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Renal function: urea, creatinina and urea nitrogen | at 48h - 28 days
  Concerning renal function at 48h after birth and in the subsequent measurements in the 7, 14, 21, 28 day of life, the values of urea, creatinine and BUN, no statistical difference was detected. Also any values outside the reference values in the high dose amino acid group was detected (Table 4).

CONTACTS AND LOCATIONS:
Overall Officials: Victor Godinez, Director, Study Director — Instituto Mexicano del Seguro Social
Locations (1):
- Instituto Mexicano del Seguro Social, León, Guanajuato, Mexico

REFERENCES:
- [Result] Moltu SJ, Blakstad EW, Strommen K, Almaas AN, Nakstad B, Ronnestad A, Braekke K, Veierod MB, Drevon CA, Iversen PO, Westerberg AC. Enhanced feeding and diminished postnatal growth failure in very-low-birth-weight infants. J Pediatr Gastroenterol Nutr. 2014 Mar;58(3):344-51. doi: 10.1097/MPG.0000000000000220. PMID 24556755
- [Result] Kotsopoulos K, Benadiba-Torch A, Cuddy A, Shah PS. Safety and efficacy of early amino acids in preterm <28 weeks gestation: prospective observational comparison. J Perinatol. 2006 Dec;26(12):749-54. doi: 10.1038/sj.jp.7211611. Epub 2006 Oct 5. PMID 17024139